CLINICAL TRIAL: NCT05734469
Title: Postoperative Recovery in Patients Undergoing Forefoot Bone Surgery. A Comparative Study of the Occurrence of a Rebound Pain Phenomenon According to the Use of Either a Popliteal Sciatic Nerve Block or a Distal Sensory Ankle Block
Brief Title: Difference in Occurrence of Rebound Pain in Patients Undergoing Surgery Under Popliteal Block or Ankle Block
Acronym: CBFR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2022/22SEP/352
Record Dates: First submitted 2023-01-17; First posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Anesthesia, Regional; Anesthesia and Analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Popliteal sciatic nerve block (Other): A local anesthetic solution of 30ml of ROPIVACAINE 0,5% (4mg/kg maximum) will be used for the popliteal sciatic nerve block (popliteal sciatic, saphenous) by real-time ultrasound guidance (associated with a standardized general anesthesia)
  Interventions: Other: Forefoot bone surgery
- Ankle block (Other): A maximum solution of 15ml of ROPIVACAINE 0. 5%( 4mg/kg maximum) for the ankle block (saphenous, superficial peroneal, deep peroneal and tibial nerves) by real-time ultrasound guidance (associated with a standardized general anesthesia)
  Interventions: Other: Forefoot bone surgery

INTERVENTIONS:
Other: Forefoot bone surgery — Elective forefoot bone surgery under popliteal sciatic nerve
  Arms: Popliteal sciatic nerve block
Other: Forefoot bone surgery — Elective forefoot bone surgery under an ankle block
  Arms: Ankle block

SUMMARY:
This is a monocentric, comparative prospective randomized controlled trial. Patients will be randomised into 2 groups and will receive either a sciatic popliteal nerve block or an ankle block (single dose locoregional block injection before the surgery) for elective forefoot surgery in addition to general anaesthesia.

The study will:

* Compare the occurrence of rebound pain and its recovery between a peripheral nerve block of the popliteal sciatic nerve and an ankle block in patients undergoing lower limb (forefoot) bone surgery under general anaesthesia combined with a PNB achieved in preoperative single injection.
* To identify the role of the type of nerve fibers anesthetized and the local inflammatory process in rebound pain development.
* Assessing the amount of the local sympathetic block induced by the locoregional anesthesia could be used a non-invasive predictive indicator of the occurrence of rebound pain depending on the nerve fibers involved (purely sensitive versus sensitive and motor).

DETAILED DESCRIPTION:
The use of peripheral nerve block (PNB) via administered local anesthetics may exacerbate the acute inflammatory process induced by surgical trauma. This exacerbation of local inflammation is a likely cause of the hyperalgesia phenomena reported upon PNB removal in the first 24 hours postoperatively. This local hyperalgesia is responsible for intense pain that is difficult to control with conventional analgesics. It is also called "rebound pain (RP)". Local anesthetics (e.g. bupivacaine) used in PNB can stimulate the expression of genes involved in inflammation and thus induce hyperalgesia following the local release of pro-inflammatory mediators (prostaglandins (prostaglandins E2 and interleukin 1β). One mechanism of action involved would be that PNB-induced increased tissue oxygen saturation ( and caused by sympathetic block associated with sensory and motor blocks). Sympathetic block and local vasodilation would promote immune cell migration at the incision site.

The primary objective will be to identify a difference in the occurrence of RP between a popliteal sciatic nerve PNB (sensory-motor block) and an ankle PNB (pure sensory block). Sensory block is currently becoming more popular because it allows for faster mobilization/functional recovery.

The secondary objective will be to identify the involvement of local sympathetic block (local vasoplegia) in the RP phenomenon. The intensity of local sympathetic block would be an indirect, non-invasive indicator of a possible modulation of local inflammation (repeated non-invasive measurement of temperature and tissue oxygen perfusion changes)

Method: Randomized patients will receive either a popliteal sciatic nerve block or an ankle block. A local anesthetic solution of 30ml of ROPIVACAINE 0. 5%,(4mg/kg maximum) will be used for popliteal sciatic nerve block (popliteal sciatic, saphenous) and a maximum solution of 15ml of ROPIVACAINE 0. 5%( 4mg/kg maximum) for ankle block (saphenous, superficial peroneal, deep peroneal and tibial nerves). Each nerve will be treated separately, anesthetized by real-time ultrasound guidance. Both groups will also receive standardized general anesthesia (induction of anesthesia by intravenous injection of Propofol, Sufentanil with maintenance of inhalation anesthesia with Sevoflurane). All patients will benefit from a standardized postoperative analgesia. The reactivation to stress of the patients will be measured perioperatively by a non-invasive monitoring of the sympathetic-parasympathetic balance (ANI, antinociception index; Metrodoloris®) based on the variability of the heart rate. The evaluation of the modulation of the local inflammation will be objectivated in an indirect way by the repeated non-invasive measurement of the modifications of temperature and tissue perfusion in oxygen (sympathetic block) at the level of the tissues close to the surgical site. The neuropathic or catastrophic nature of the pain as well as the preoperative anxiety will be collected by means of specific questionnaires (APAIS /Catastrophisation /CSI..). Patients will be discharged from the hospital on day 1 or day 2 postoperatively with a standardized analgesic treatment. Under the close coordination of the investigating physician, the monitoring of the patients' postoperative pain will be done from the PACU with the participation of the recovery room nursing team, but also by the Pops pain team during their brief period of hospitalization on the floor. Patients will be discharged from the hospital on postoperative day 1 or 2 with standardized analgesic treatment. On their return home, the patients will be followed up by telephone calls (investigating physician), according to the study protocol established at D4 D30 and at 3 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Any surgery of the bones of the lower limbs performed as part of a PNB associated with general anaesthesia after lower limb bone surgery
* Patient aged between 18 and 75 years old.

Exclusion Criteria:

* refusal to participate
* contraindication to the use of local anesthetics
* contraindication to the use of general anesthesia
* contraindication to regular use of postoperative analgesics like non-steroidal anti-inflammatory drugs and paracetamol
* cognitive disorders
* inability to answer perioperative questionnaires (language problem).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-02-15 (Estimated); Primary Completion 2024-02-15 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Difference in the occurrence of rebound pain according to the type of PNB | Through study completion, an average of 1 year
  The investigators wished to prospectively evaluate and compare the incidence of the occurrence of RP, in the context of popliteal sciatic nerve PNB (sensory-motor block) and in the context of distal ankle PNB (pure sensory block). RP was defined in this study as severe pain with a Numerating Rating Scale of Spasticity (NRS) score ≥ 7/10 within the first 24 hours after performing the PNB.

SECONDARY OUTCOMES:
The importance of the local sympathetic block induced by the locoregional anesthesia as well as the type of anesthetized nerve fibers in the rebound pain process. | Through study completion, an average of 1 year
  The investigators are interested in assessing the impact of sympathetic fibre block, thus the degree of local vasoplegia, on the incidence of the RP phenomenon. Sympathetic block (indirect indicator of modulation and increase of local inflammation) will be assessed by:
  * Repeated non-invasive measurement of local temperature changes (Digital infrared thermometer in the degree Celsius),
  * Tissue oxygen perfusion by Periflux 6000 (oxygen values transcutaneous in millimeters of mercury ) and by the INVOS™ system, which monitors real-time changes in the percentage of regional oxygen saturation (rSO2) of blood in body tissues below the sensor.
  * Measurement of inflammatory mediators by blood analysis, C-Réactive Proteine (CRP) value (in milligrams/liter) and NLR value (neutrophil to lymphocyte ratio).
Predictors of Pain Rebound in the Context of Forefoot Surgery with BNP | Through study completion, an average of 1 year
  Preoperative questionnaires will be completed by the patients to identify possible predictive factors for the occurrence of RP and thus determine profiles more at risk. For this purpose, each patient will have to complete preoperatively :
  * A questionnaire assessing catastrophization which includes the evaluation of rumination , amplification , and helplessness (13 items scored from 0 to 4)
  * A questionnaire assessing preoperative anesthetic and surgical anxiety APAIS (Amsterdam Preoperative Anxiety and Information Scale). The score can range from 6 ("no anxiety") to 30 ("very anxious").
  * A questionnaire evaluating the central sensitivity CSI (Central Sensitization Index) (9 questions)
  * The DN4 (4 questions) and DN2 (2 questions) questionnaires which will allow to evaluate the risk of developing neuropathic pain .

CONTACTS AND LOCATIONS:
Overall Officials: Nassim TOUIL, MD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barry GS, Bailey JG, Sardinha J, Brousseau P, Uppal V. Factors associated with rebound pain after peripheral nerve block for ambulatory surgery. Br J Anaesth. 2021 Apr;126(4):862-871. doi: 10.1016/j.bja.2020.10.035. Epub 2020 Dec 31. PMID 33390261
- [Background] Streb T, Schneider A, Wiesmann T, Riecke J, Schubert AK, Dinges HC, Volberg C. [Rebound pain-From definition to treatment]. Anaesthesiologie. 2022 Aug;71(8):638-645. doi: 10.1007/s00101-022-01120-z. Epub 2022 May 5. German. PMID 35513729
- [Background] Hamilton DL. Rebound pain: distinct pain phenomenon or nonentity? Br J Anaesth. 2021 Apr;126(4):761-763. doi: 10.1016/j.bja.2020.12.034. Epub 2021 Feb 5. No abstract available. PMID 33551124
- [Background] Touil N, Pavlopoulou A, Barbier O, Libouton X, Lavand'homme P. Evaluation of intraoperative ketamine on the prevention of severe rebound pain upon cessation of peripheral nerve block: a prospective randomised, double-blind, placebo-controlled study. Br J Anaesth. 2022 Apr;128(4):734-741. doi: 10.1016/j.bja.2021.11.043. Epub 2022 Feb 23. PMID 35219449
- [Background] Sort R, Brorson S, Gogenur I, Nielsen JK, Moller AM. Rebound pain following peripheral nerve block anaesthesia in acute ankle fracture surgery: An exploratory pilot study. Acta Anaesthesiol Scand. 2019 Mar;63(3):396-402. doi: 10.1111/aas.13290. Epub 2018 Nov 8. PMID 30411313
- [Background] Sort R, Brorson S, Gogenur I, Hald LL, Nielsen JK, Salling N, Hougaard S, Foss NB, Tengberg PT, Klausen TW, Moller AM. Peripheral nerve block anaesthesia and postoperative pain in acute ankle fracture surgery: the AnAnkle randomised trial. Br J Anaesth. 2021 Apr;126(4):881-888. doi: 10.1016/j.bja.2020.12.037. Epub 2021 Feb 2. PMID 33546844
- [Background] Jen TTH, Ke JXC, Wing KJ, Denomme J, McIsaac DI, Huang SC, Ree RM, Prabhakar C, Schwarz SKW, Yarnold CH. Development and internal validation of a multivariable risk prediction model for severe rebound pain after foot and ankle surgery involving single-shot popliteal sciatic nerve block. Br J Anaesth. 2022 Jul;129(1):127-135. doi: 10.1016/j.bja.2022.03.030. Epub 2022 May 12. PMID 35568510
- [Background] Goldstein RY, Montero N, Jain SK, Egol KA, Tejwani NC. Efficacy of popliteal block in postoperative pain control after ankle fracture fixation: a prospective randomized study. J Orthop Trauma. 2012 Oct;26(10):557-61. doi: 10.1097/BOT.0b013e3182638b25. PMID 22732860
- [Background] Yamada T, Hasegawa-Moriyama M, Kurimoto T, Saito T, Kuwaki T, Kanmura Y. Peripheral Nerve Block Facilitates Acute Inflammatory Responses Induced by Surgical Incision in Mice. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):593-600. doi: 10.1097/AAP.0000000000000458. PMID 27547899
- [Background] Tighe PJ, Elliott CE, Lucas SD, Boezaart AP. Noninvasive tissue oxygen saturation determined by near-infrared spectroscopy following peripheral nerve block. Acta Anaesthesiol Scand. 2011 Nov;55(10):1239-46. doi: 10.1111/j.1399-6576.2011.02533.x. Epub 2011 Sep 26. PMID 22092129